CLINICAL TRIAL: NCT00891319
Title: Contralaterally Controlled FES for Chronic Arm/Hand Hemiplegia: Single-Site RCT
Brief Title: Electrical Stimulation for Recovery of Hand Function in Chronic Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Jayme Knutson, Assistant Professor, Physical Medicine and Rehabilitation, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD059814 (NIH); R01HD059814 (NIH)
Record Dates: First submitted 2008-09-25; First posted 2009-05-01 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Stroke; Hemiparesis; Hemiplegia
Keywords: hand; stroke; hemiplegia; electrical stimulation; recovery
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- CCFES (Experimental): CCFES - Contralaterally Controlled Functional Electrical Stimulation
  * Electrical stimulator
  * Stimulation to finger and thumb extensors only in response to, and with an intensity proportional to, opening of the contralateral unimpaired hand.
  * A glove instrumented with sensors and worn on the unimpaired hand detects the degree of hand opening and determines stimulation intensity.
  * Therapy sessions are done with the subject being assisted by the CCFES system.
  Interventions: Device: Electrical stimulator
- cNMES (Active Comparator): cNMES - Cyclic NeuroMuscular Electrical Stimulation
  * Electrical stimulator
  * Preprogrammed cycles of finger and thumb extensor stimulation repeatedly and automatically open the hand.
  * Subject instructed to not move the contralateral arm/hand during stimulation.
  * Therapy sessions are done without the stimulation system.
  Interventions: Device: Electrical stimulator

INTERVENTIONS:
Device: Electrical stimulator — • 12-week intervention
  1. Therapist-guided task practice performed twice a week in the research laboratory. (Device used for CCFES group but not for cNMES group during these sessions.)
  2. Self-administered CCFES or cNMES-mediated hand opening exercise performed 10 sessions per week at home.

SUMMARY:
Impaired hand function is one of the most frequently persisting consequences of stroke. The purpose of this study is to compare two different treatments -- Contralataterally Controlled Functional Electrical Stimulation (CCFES) and Cyclic Neuromuscular Electrical Stimulation (cNMES) -- for improved recovery of hand function after stroke.

DETAILED DESCRIPTION:
Hemiparesis of the upper limb is one of the most serious and most common impairments resulting from stroke. Approximately 75% of the over 750,000 strokes that occur annually in the United States cause some degree of upper extremity paralysis. Approximately 65% of stroke survivors still cannot use their affected hand to assist with activities of daily living 6 months after their stroke. The impact of upper extremity impairments on disability and health is great, yet there are relatively few rehabilitation interventions designed to restore function to the impaired upper limb. Therefore, our long-term objective is to develop upper extremity rehabilitation therapies that are effective at restoring arm and hand function, that are applicable across a wide range of impairment severity, and that are readily implemented in the present healthcare environment.

The purpose of this study is to estimate the efficacy of Contralataterally Controlled Functional Electrical Stimulation (CCFES) in reducing upper extremity impairment and activity limitation in chronic upper extremity hemiplegia. CCFES is a rehabilitation intervention in which neuromuscular electrical stimulation (NMES) is applied to the finger and thumb extensor muscles of the paretic upper limb to open the hand. The stroke survivor controls the stimulation intensity, and consequent degree of hand opening, by modulating the degree of opening of the contralateral unimpaired hand, which is detected by an instrumented glove. Thus, volitional opening of the unaffected hand produces stimulated opening of the affected hand. The stimulation paradigm is used to assist the stroke survivor in practicing functional tasks with their affected hand. We will conduct a randomized controlled trial in which chronic stroke survivors (>6 months post-stroke) will be randomly assigned to receive 12 weeks of CCFES or cyclic NMES, an intervention that provides electrical stimulation of the hand extensors, but with preprogrammed timing and intensity. Randomization will be stratified on two levels of baseline hand impairment defined by the degree of voluntary finger extension present. Assessments of upper extremity impairment and activity limitation will be made every 3 weeks during the treatment period and every 2 months during a 6-month follow-up period.

This study is the first randomized controlled trial of CCFES in chronic upper extremity hemiplegia. Ultimately, the information learned in this study will serve to accelerate the development of treatments for reducing post-stroke disability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* > 6 months of first hemorrhagic or nonhemorrhagic stroke
* Able to recall 2 of 3 items after 30 minutes
* MRC ≤ 4 for finger extensors on paretic side
* Able to follow 3-stage commands
* Functional movement of shoulder and elbow (e.g., can reach ¾ hand-to- mouth movement) of paretic side
* Caregiver available to assist with device and compliance if needed
* Skin intact on hemiparetic arm
* Medically stable
* Surface NMES trial opens hand without pain
* Full volitional hand opening/closing of contralateral hand
* Upper extremity hand section of FMA < 11/14
* Able to hear and respond to stimulator/cue box auditory cues
* Completed occupational therapy (no concomitant OT)

Exclusion Criteria:

* Lack of functional PROM of the wrist or fingers of affected side
* Severe shoulder or hand pain (unable to position hand in the workspace without pain)
* Uncontrolled seizure disorder
* Insensate forearm and/or hand
* Uncompensated hemi-neglect (extinguishing to double simultaneous stimulation)
* Edema of the affected forearm and/or hand
* History of cardiac arrhythmias with hemodynamic instability
* Cardiac pacemaker or other implanted electronic system
* Pregnant
* IM Botox injections in any UE muscle in the last 3 months
* Parkinson's disease, SCI, TBI, or MS
* Ipsilateral motor neuron lesion

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jayme S. Knutson, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knutson JS, Harley MY, Hisel TZ, Chae J. Improving hand function in stroke survivors: a pilot study of contralaterally controlled functional electric stimulation in chronic hemiplegia. Arch Phys Med Rehabil. 2007 Apr;88(4):513-20. doi: 10.1016/j.apmr.2007.01.003. PMID 17398254
- [Background] Glanz M, Klawansky S, Stason W, Berkey C, Chalmers TC. Functional electrostimulation in poststroke rehabilitation: a meta-analysis of the randomized controlled trials. Arch Phys Med Rehabil. 1996 Jun;77(6):549-53. doi: 10.1016/s0003-9993(96)90293-2. PMID 8831470
- [Background] Chae J, Bethoux F, Bohine T, Dobos L, Davis T, Friedl A. Neuromuscular stimulation for upper extremity motor and functional recovery in acute hemiplegia. Stroke. 1998 May;29(5):975-9. doi: 10.1161/01.str.29.5.975. PMID 9596245
- [Background] Luft AR, McCombe-Waller S, Whitall J, Forrester LW, Macko R, Sorkin JD, Schulz JB, Goldberg AP, Hanley DF. Repetitive bilateral arm training and motor cortex activation in chronic stroke: a randomized controlled trial. JAMA. 2004 Oct 20;292(15):1853-61. doi: 10.1001/jama.292.15.1853. PMID 15494583
- [Background] Whitall J, McCombe Waller S, Silver KH, Macko RF. Repetitive bilateral arm training with rhythmic auditory cueing improves motor function in chronic hemiparetic stroke. Stroke. 2000 Oct;31(10):2390-5. doi: 10.1161/01.str.31.10.2390. PMID 11022069
- [Background] Mudie MH, Matyas TA. Can simultaneous bilateral movement involve the undamaged hemisphere in reconstruction of neural networks damaged by stroke? Disabil Rehabil. 2000 Jan 10-20;22(1-2):23-37. doi: 10.1080/096382800297097. PMID 10661755
- [Derived] Knutson JS, Gunzler DD, Wilson RD, Chae J. Contralaterally Controlled Functional Electrical Stimulation Improves Hand Dexterity in Chronic Hemiparesis: A Randomized Trial. Stroke. 2016 Oct;47(10):2596-602. doi: 10.1161/STROKEAHA.116.013791. Epub 2016 Sep 8. PMID 27608819
- See also: Cleveland FES Center — http://fescenter.org/index.php
- See also: The MetroHealth System - Clinical Trials — http://www.metrohealth.org/body.cfm?id=2438

RESULTS

PARTICIPANT FLOW:
Groups:
- CCFES: CCFES - Contralaterally Controlled Functional Electrical Stimulation
  *Stimulation to paretic finger and thumb extensors only in response to, and with an intensity proportional to, opening of the contralateral unimpaired hand. A glove instrumented with sensors and worn on the unimpaired hand detects the degree of hand opening and controls stimulation intensity delivered to the affected hand.
  12-week intervention
  1. Lab: Therapist-guided CCFES-assisted task practice performed twice a week in the research laboratory.
  2. Home: Self-administered CCFES-mediated hand opening exercise performed 10 sessions per week at home.
- cNMES: cNMES - Cyclic NeuroMuscular Electrical Stimulation
  *Preprogrammed cycles of finger and thumb extensor stimulation repeatedly and automatically open the paretic hand.
  12-week intervention
  1. Lab: Therapist-guided task practice performed twice a week in the research laboratory.
  2. Home: Self-administered cNMES-mediated hand opening exercise performed t10 sessions per week at home.
Period: Overall Study
Arm/Group | CCFES | cNMES
Started | 40 | 40
Completed | 32 | 40
Not Completed | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CCFES | cNMES | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55.4 [48.1 to 66.2] | 56.3 [51.9 to 65.2] | 56.2 [51.0 to 65.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 26 | 25 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 17 | 39
  White | 18 | 23 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Years Since Stroke [Median (Inter-Quartile Range); unit: years since stroke] | 1.8 [0.8 to 3.5] | 1.6 [1.0 to 6.0] | 1.6 [0.9 to 4.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in Box and Block Test Score at 6 Mo Post-Treatment
Description: The Box and Blocks test counts how many times the participant can pick up 1 block at t time, move it over a partition, and release it in a target area within 60 seconds.
  The minimum score is 0. There is no maximum score. The average score of healthy individuals within the age range of this study ranges from 70 to 79.
  Higher scores are considered to be a better outcome. For each individual, the score prior to treatment was subtracted from the score at 6 months after completion of treatment. Then for each treatment group, these change scores were averaged.
Time Frame: 2 timepoints: Prior to treatment, and 6 months after completion of treatment.
Measure: Mean (95% Confidence Interval); unit: blocks
Groups:
- cNMES: cNMES - Cyclic NeuroMuscular Electrical Stimulation
  *Preprogrammed cycles of finger and thumb extensor stimulation repeatedly and automatically open the paretic hand.
  12-week intervention
  1. Lab: Therapist-guided task practice performed twice a week in the research laboratory.
  2. Home: Self-administered cNMES-mediated hand opening exercise performed 10 sessions per week at home.
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 32 | 40
blocks | 4.6 [2.2 to 7.0] | 1.8 [0.6 to 3.0]

2. Secondary Outcome: Change in Arm Motor Abilities Test Score at 6-Month Post-Treatment
Description: The Arm Motor Abilities Test assesses the participant's ability to execute specific upper limb tasks and does not allow for compensation with the unimpaired side. The test consists of 9 compound tasks composed of 1 to 3 component tasks, each of which is rated on a 0 - 5 ordinal scale: 0, no attempt to use affected limb; 1, attempt to use affected limb but it does not participate functionally; 2, affected limb is used only as a helper or stabilizer; 3, affected limb is used slowly or within synergy patterns; 4, almost normal use of affected limb; 5, normal use. The final score is the average of all component task scores across all 9 compound tasks.
  The minimum score is 0; maximum score is 5. Higher scores are considered to be a better outcome. For each individual, the score prior to treatment was subtracted from the score at 6 months after completion of treatment. Then for each treatment group, these change scores were averaged.
Time Frame: 2 timepoints: Prior to treatment, and 6 months after completion of treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 32 | 40
units on a scale | 0.18 [0.06 to 0.31] | 0.04 [-0.07 to 0.15]

3. Secondary Outcome: Change in Upper Extremity Fugl-Meyer Score at 6-Months Post-Treatment
Description: The Upper Extremity Fugl-Meyer (UEFM) Assessment is a measure of upper limb motor impairment. Participants are asked to attempt to perform a list of very specific movements of the arm, elbow, forearm, wrist, and hand that take into account synergy patterns, isolated strength, coordination, and hypertonia. Each movement attempt is graded on a 3-point ordinal scale (0, cannot perform; 1, perform partially; and 2, perform fully) and these subscores are summed to provide a maximum score of 66, minimum score of 0.
  Higher scores are considered to be a better outcome. For each individual, the score prior to treatment was subtracted from the score at 6 months after completion of treatment. Then for each treatment group, these change scores were averaged.
Time Frame: 2 timepoints: Prior to treatment, and 6 months after completion of treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CCFES | cNMES
Number analyzed (Participants) | 32 | 40
units on a scale | 2.4 [0.5 to 4.3] | 2.2 [0.7 to 3.7]

ADVERSE EVENTS:
Arm/Group | CCFES | cNMES
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 4/40 | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CCFES (N=40) | cNMES (N=40)
Headaches after therapy sessions (General disorders) | 1 | 0
Skin irritation from electrodes (Skin and subcutaneous tissue disorders) | 2 | 1
Stimulation uncomfortable (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes